CLINICAL TRIAL: NCT01875783
Title: Diabetic Macular Edema Found by OCT Utilization at Non-ophthalmic Diabetes Care Visits
Brief Title: OCT Screening for Diabetic Macular Edema at Primary Diabetes Care Visits
Acronym: DME FOUND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Genentech, Inc. (Industry); Juvenile Diabetes Research Foundation (Other); Optovue (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2011-17
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Results first posted 2017-09-20 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Diabetes; Diabetic Macular Edema; Diabetic Retinopathy
Keywords: diabetes; diabetic macular edema; diabetic retinopathy; optical coherence tomography
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Primary diabetes care specialists masked to results of OCT intervention
Oversight: Data Monitoring Committee: No

ARMS (1):
- OCT imaging (Experimental): All study participants will undergo optical coherence tomography imaging and will be referred to a retina specialist for further standard care evaluation and management if they are identified as having diabetic macular edema or the scan quality is not sufficient to evaluate macular status.
  Interventions: Device: OCT imaging

INTERVENTIONS:
Device: OCT imaging — Optical coherence tomography (OCT) imaging is a noninvasive, rapid, and readily performed method for evaluating the anatomy of the central retina.

SUMMARY:
The purpose of this protocol is to determine whether point of care optical coherence tomography (OCT) imaging combined with an OCT-guided retinal referral algorithm at primary diabetes care visits increases rates of retina specialist eye care for patients with diabetic macular edema. The hypothesis is that OCT imaging with an automated OCT-guided referral algorithm will enable identification of patients at risk for vision loss from diabetic macular edema and facilitate direct referral to retina specialists for more timely evaluation and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes mellitus as evidenced by:
* Current regular use of insulin or oral anti-hyperglycemia agents for the treatment of diabetes OR
* Documented diabetes by American Diabetes Association and/or World Health Organization criteria
* Age greater than or equal to 18 years old
* Diabetes duration of 10 more years OR last measured HbA1c of 10% or more
* Able and willing to participate in study procedures and comply with study follow-up visits
* Able to give informed consent for study participation
* Not moving out of the study area during the 1 year follow-up period

Exclusion Criteria:

* Unable to cooperate with the OCT image acquisition procedure or other study procedures
* Unable or unwilling to comply with the study follow-up visits
* Unable or unwilling to sign form for release of retinal medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2014-03-17 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2016-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K Sun, MD, Principal Investigator — Joslin Diabetes Center
Locations (4):
- United States (4):
  - Joslin Diabetes Center, Boston, Massachusetts
  - OuterCape Health Services, Inc, Wellfleet, Massachusetts
  - SUNY Upstate Medical University, Syracuse, New York
  - University of Endocrine Consultants, Chattanooga, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OCT Imaging
Started | 385
Completed | 385
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OCT Imaging
Number analyzed (Participants) | 385
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 294
  >=65 years | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 193
  Male | 192
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 385

OUTCOME MEASURES:

1. Primary Outcome: Rates of Retina Care Referral for Patients With Diabetic Macular Edema
Description: Percentage of participants who are referred to a retina specialist for evaluation and management of DME after OCT imaging and OCT-guided referral algorithm
Time Frame: Baseline visit
Measure: Count of Participants; unit: Participants
Groups:
- Retina Specialist Care: Percentage of participants who follow-up with a retina specialist for evaluation and management of DME after OCT imaging and OCT-guided referral algorithm as compared with the percentage of patients currently receiving retina eye care (assessed by study participant self-report as well as by determination of historical retina eye care rates from documentation in the medical records of study-eligible patients seen within the previous 6 months)
Arm/Group | Retina Specialist Care
Number analyzed (Participants) | 385
Participants | 44

2. Secondary Outcome: Retinal Referral Rates for Patients With DME
Description: Count of eyes that are referred to a retina specialist for evaluation and management of DME after OCT imaging and OCT-guided referral algorithm
Time Frame: Baseline visit
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Groups:
- Eyes That Have Undergone OCT Imaging: All study participants will undergo optical coherence tomography imaging and will be referred to a retina specialist for further standard care evaluation and management if they are identified as having diabetic macular edema or the scan quality is not sufficient to evaluate macular status.
  OCT imaging: Optical coherence tomography (OCT) imaging is a noninvasive, rapid, and readily performed method for evaluating the anatomy of the central retina.
Arm/Group | Eyes That Have Undergone OCT Imaging
Number analyzed (Participants) | 385
Number analyzed (eyes) | 761
eyes | 59

3. Secondary Outcome: Rates of Retinal Treatment for Patients With DME
Description: Percentage of participants are referred by OCT-guided algorithm who are confirmed to have vision threatening retinopathy at first visit with retina specialist after study enrollment
Time Frame: One month
Population: This is the subgroup of participants who were referred for retinal care by the OCT guided referral algorithm
Measure: Count of Participants; unit: Participants
Groups:
- Participants Referred for Retina Care: Study participants identified for retina referral by the OCT guided referral algorithm.
Arm/Group | Participants Referred for Retina Care
Number analyzed (Participants) | 34
Participants | 14

4. Secondary Outcome: Rates of Retinal Treatment Over 1 Year for Patients With DME
Description: Percentage of participants who are referred by OCT guided algorithm to a retina specialist who receive treatment for DME over the course of 9 months follow-up by retina specialist
Time Frame: 9 months
Population: This is the subgroup of participants who were referred for retina care by the OCT guided referral algorithm.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Referred for Retina Care
Number analyzed (Participants) | 34
Participants | 18

ADVERSE EVENTS:
Arm/Group | OCT Imaging
All-Cause Mortality (participants affected / at risk) | 0/385
Serious Adverse Events (participants affected / at risk) | 0/385
Other Adverse Events (participants affected / at risk) | 0/385

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No